CLINICAL TRIAL: NCT03589443
Title: Phase I In-vivo Study of Multiplexed Heptapeptides for Detection of Neoplasia in the Esophagus
Brief Title: Study of Multiplexed Heptapeptides for Detection of Neoplasia in the Esophagus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Danielle Kim Turgeon, Professor of Internal Medicine, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00137993
Record Dates: First submitted 2018-06-21; First posted 2018-07-17 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Multiplexed heptapeptides (Experimental): QRH & KSP sprayed onto area of interest and imaged before and after application
  Interventions: Drug: Multiplexed heptapeptides

INTERVENTIONS:
Drug: Multiplexed heptapeptides — Heptapeptides QRH and KSP

SUMMARY:
The overall aim of this feasibility study is to develop new technologies for improved detection of Barrett's neoplasia using the scanning fiber endoscope(SFE) multiplexed imaging system. This study will combine the use of fluorescent-labeled peptides that bind specifically to pre-cancerous mucosa in the esophagus for use as novel imaging agents to guide endoscopic biopsy or endoscopic mucosal resection (EMR). This Phase 1 study will be used to provide early evidence of efficacy for the topical application of a panel of two peptides that bind to molecular targets that are specific for esophageal dysplasia. A panel is needed because cancer in the esophagus is genetically heterogeneous. The study will look at peptide binding in subjects with known or suspected Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected Barrett's esophagus
* Scheduled for a clinically-indicated upper endoscopy
* Medically cleared for the procedure
* Willing and able to sign informed consent

Exclusion Criteria:

* Known allergy or negative reaction to the near infrared fluorophores Cy5, li-cor IRDye800CW, or derivatives
* One active chemotherapy or radiation treatment
* Pregnant or trying to conceive

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Validate the binding of the peptides using the SFE | 1 year
  The binding of the fluorescent-labeled peptides (QRH-882260 and KSP-910638G) that bind to EGFR and HER2 using an SFE molecular imaging system (SFE) determined using the tumor-to-background ratio for fluorescence intensities

SECONDARY OUTCOMES:
Use of the SFE to detect QRH and KSP via signal to noise ratio (SNR) | 1 year
  One aspect of feasibility will be shown by examining the SNR of the images collected.
Use of the SFE to detect QRH and KSP via tumor-to-background ratio | 1 year
  One aspect of feasibility will be shown by examining the tumor-to-background ratio of the images collected.
Use of the SFE to detect QRH and KSP via contrast | 1 year
  One aspect of feasibility will be shown by examining the contrast in the two channels in the images collected.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States